CLINICAL TRIAL: NCT02627820
Title: An 18 Month Open Label Study Of The Tolerability And Efficacy Of An Antisense Oligonucleotide In Patients With Wild-Type Transthyretin Amyloid Cardiomyopathy (Senile Systemic Amyloidosis)
Brief Title: The Effect of an Antisense Oligonucleotide to Lower Transthyretin (TTR) Levels on the Progression of -Wild-type TTR Involving the Heart
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry); Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Rodney H. Falk, MD, Director, Brigham and Women's Cardiac Amyloidosis Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-P001574
Record Dates: First submitted 2015-11-19; First posted 2015-12-11 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-01

CONDITIONS: Amyloidosis
Keywords: Senile; ATTRwt; wild-type transthyretin amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Oligonucleotides, Antisense

ARMS (1):
- Experimental Drug (Experimental): Isis 420915/GSK 299872, an antisense oligonucleotide. Administered subcutaneously three times per week for the first week, and then weekly for 18 months. Each dose shall contain 300 mg of active drug.
  Interventions: Drug: Isis 420915/GSK 299872

INTERVENTIONS:
Drug: Isis 420915/GSK 299872 — Open label study in comparison to historic control.
  Other Names: Antisense oligonucleotide

SUMMARY:
ATTRwt (also known as senile systemic, or senile cardiac amyloidosis) is a progressive heart disease, causing congestive heart failure. It is caused by amyloid protein deposits in the heart, that are derived from a normal protein, TTR, made in the liver. The aim of the study is to determine whether lowering the blood levels of TTR, by a weekly injection of a compound designed specifically to do this, will slow the progression of the disease when treated patients are compared to previously-followed patients who were not receiving this drug. The study also aims to determine how well this drug is tolerated and the existence and severity of any drug side-effects.

ELIGIBILITY:
All patients with documented SSA will be considered for inclusion. SSA is defined as an echocardiographic appearance of left ventricular wall thickness of 13 mm or more, in the absence of uncontrolled hypertension, and with a positive biopsy for amyloid, which also stains positive for TTR by immunochemistry or mass spectrometry. For the definition of SSA, genetic testing should be negative for a mutation. Identification of amyloid type is standard of care for all patients seen at the Cardiac Amyloidosis Program and the presence of a clinically -obtained positive biopsy will be a requirement for study inclusion. The positive biopsy can be from any organ, providing that the echocardiographic appearance is typical of amyloidosis.

Inclusion Criteria:

1. Patients should, in the opinion of the Investigator, be in a stable state in terms of NYHA class. Class I-III patients will be recruited.
2. Age 50-90 years
3. Male or non-pregnant, non-lactating females. If a woman is premenopausal, or a male partners with a premenopausal woman, she/he must be willing to use the following methods of contraception: condoms, oral/hormonal contraception, Intrauterine Device, diaphragm, or abstinence
4. Written informed consent to be obtained prior to study treatment
5. Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens
6. Molecular definition of the absence of a TTR mutation or immunohistochemical staining of amyloid fibrils with anti TTR antibody and negative genetic testing for a TTR mutation.
7. Willingness to return to the treating center for follow-up.
8. Willingness and ability to self-administer, or to have spouse administer weekly subcutaneous injections of study drug.

Exclusion Criteria:

1. Patients who, in the opinion of the Investigator, require further adjustment of diuretics at the time of screening to achieve optimal treatment of heart failure. Once stable for 2 weeks, patients in Class I-III will become eligible for inclusion.
2. Patients with NYHA class 4 congestive heart failure.
3. Concomitant non-amyloid heart disease that might, in the opinion of the investigator, cause changes in strain imaging on serial follow-up (e.g. aortic stenosis of greater than mild severity, unstable coronary artery disease).
4. Prior liver transplantation or liver transplantation anticipated in less than 6 months;
5. ALT and/or AST ³ 2 x ULN and/or Alkaline phosphatase ³ 2 x UNL;
6. Estimated glomerular filtration rate (EGFR) < 50 ml/min;
7. Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study;
8. History of poor compliance with medications or medical treatment, based on a review of medical records.
9. History of hypersensitivity to any of the ingredients of the study therapy;
10. Use of any investigational drug for amyloidosis within 4 weeks prior to study entry or during the study.
11. Current use of tafamidis, diflunisal, doxycycline or TUDCA for therapy of amyloidosis.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Systolic strain imaging by echocardiographic speckle tracking | Month 12
  The primary echocardiographic parameter to be measured will be longitudinal left ventricular (LV) strain (units = % LV longitudinal shortening) as compared to baseline.

SECONDARY OUTCOMES:
Systolic strain evaluation by echocardiography | Secondary analysis will occur at 18 months
  The primary echocardiographic parameter measured will be longitudinal left ventricular (LV) strain (units = %).
Echocardiographic determination of Mean thickness of LV septum and posterior wall (units = mm) | 12 months
Echocardiographic determination of Mean thickness of LV septum and posterior wall (units = mm) | 18 months
Echocardiographic determination of LV ejection fraction (units = %) | 12 months
Echocardiographic determination of LV ejection fraction (units = %) | 18 months
LV mass measurement by Cardiac MRI (cMRI) (units = grams) | 18 months
LV cellular component as determined by cMRI (units = % of total LV mass) | 12 months
LV cellular component as determined by cMRI (units = % of total LV mass) | 18 months
LV extracellular component as determined by cMRI (units = % of total LV mass) | 12 months
LV extracellular component as determined by cMRI (units = % of total LV mass) | 18 months
Extent of cMRI late gadolinium enhancement of the LV (unites = % of area) | 12 months
Extent of cMRI late gadolinium enhancement of the LV (unites = % of area) | 18 months
LV mass measurement by Cardiac MRI (cMRI) (units = grams) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Falk, MD, Principal Investigator — Brigham and Women's Hospital